CLINICAL TRIAL: NCT01731041
Title: Impact of Ticagrelor Re-load on Pharmacodynamic Profiles in Patients on Maintenance Ticagrelor Therapy
Brief Title: Impact of Ticagrelor Re-load on Pharmacodynamic Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFJ 2012-096
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary disease, platelet function, platelet inhibitors
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor 180mg (Experimental): Patients randomized to this arm will be administered 180 mg of ticagrelor (experimental arm, loading dose).
  Interventions: Drug: Ticagrelor 180mg
- Ticagrelor 90mg (Active Comparator): Patients randomized to this arm will be administered 90 mg dose of ticagrelor (active comparator, standard dose).
  Interventions: Drug: Ticagrelor 90mg

INTERVENTIONS:
Drug: Ticagrelor 180mg — Patients will receive 180 mg of ticagrelor
  Other Names: Brilinta
  Arms: Ticagrelor 180mg
Drug: Ticagrelor 90mg — Patients will receive 90 mg of ticagrelor
  Other Names: Brilinta
  Arms: Ticagrelor 90mg

SUMMARY:
Platelets are parts of your blood that stick together to help form a clot. The stickier your platelets are, the greater your chance of having a heart attack. A clot in the wrong place can lead to a heart attack or stroke. Ticagrelor (Brilinta) keeps platelets from sticking together and it helps people from having a heart attack. The American College of Cardiology has recommended a combination of aspirin and Brilinta as one of the best treatments for the prevention of heart attacks, and death in patients who have had a heart attack or coronary stents. However, it is unknown if Brilinta may improve its work to keep platelets from sticking together giving a loading dose in patients already treated with Brilinta. A loading dose is a one-time increased dose of the same drug. The purpose of this study is to demonstrate whether the platelets of patients treated with Brilinta become less sticky when Brilinta is re-loaded.

DETAILED DESCRIPTION:
A higher degree of platelet inhibition remains the goal of peri-interventional and long-term anti-thrombotic therapy in patients with coronary artery disease. Previous observations have shown that in patients on clopidogrel therapy undergoing percutanoues coronary intervention who get re-loaded with clopidogrel obtain enhanced platelet inhibition. Ticagrelor represents a new class of nonthienopyridine platelet inhibitors designed to address the limitations of current oral antiplatelet therapy, which has been recently approved for clinical use. However, to date it is unknown if greater inhibition of platelet aggregation can be achieved by adding a ticagrelor loading dose in patients already on maintenance ticagrelor therapy (90 mg twice daily). In addition, how to manage patients undergoing coronary interventions already on chronic ticagrelor therapy with regards to ticagrelor loading is an emerging clinical question which has yet to be explored. Therefore, understanding the pharmacodynamic implications of a ticagrelor re-load strategy in patients on already on chronic ticagrelor therapy is warranted. The scope of the present study is to evaluate the impact of ticagrelor re-load in patients on chronic ticagrelor therapy. A total of 60 patients will be randomized into one of the following two arms of treatment: 1) 90 mg of ticagrelor; 2) 180 mg of ticagrelor. Pharmacodynamic assessments will be performed at baseline, 1-hour and 4-hour after dosing administration. Comparison between baseline and 4-hour values in term of platelet P2Y12 reactivity index determined by whole blood vasodilator-stimulated phosphoprotein will be the primary end-point of the study. Secondary endpoints will include other pharmacodynamic measures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical indication to be on ticagrelor therapy (90mg/bid)
2. On treatment with ticagrelor 90mg twice daily for at least 14 days
3. Age between 18 to 80 years
4. On aspirin <100mg/day

Exclusion Criteria:

1. History of intracranial bleeding
2. Severe hepatic impairment (ALT >2.5 times the upper limit of normal)
3. Active bleeding or propensity to bleed
4. Recent antiplatelet treatment (< 14 days) with a glycoprotein IIb/IIIa antagonist

6. Platelet count <80x106/mL 7. Hemodynamic instability 8. Serum creatinine <30 mL/min 9. On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban) 10. Patients with sick sinus syndrome or II or III degree AV block without pacemaker protection 12. Drugs interfering CYP3A4 metabolism (to avoid interaction with Ticagrelor): ketoconazole, itraconazole, voriconazole, clarithromicin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir and telithromizycin 13. Hemoglobin < 10g/dL 14. Pregnant females [women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study].

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Cho JR, Rollini F, Franchi F, DeGroat C, Bhatti M, Dunn EC, Ferrante E, Muniz-Lozano A, Suryadevara S, Zenni MM, Guzman LA, Bass TA, Angiolillo DJ. Pharmacodynamic Effects of Ticagrelor Dosing Regimens in Patients on Maintenance Ticagrelor Therapy: Results From a Prospective, Randomized, Double-Blind Investigation. JACC Cardiovasc Interv. 2015 Jul;8(8):1075-1083. doi: 10.1016/j.jcin.2015.02.022. Epub 2015 Jun 24. PMID 26117466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened at the Division of Cardiology of the University Of Florida College Of Medicine - Jacksonville
Groups:
- Ticagrelor 180mg; Ticagrelor 90mg: A total of 60 subjects will be included in this study and will be randomized in a prospective, double-blind fashion in two treatment groups: 1) 90 mg dose of ticagrelor (active comparator, standard dose); 2) 180 mg of ticagrelor (experimatal arm, loading dose).
Period: Overall Study
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients had experienced an ACS and had a guideline-based indication to be on DAPT with aspirin and ticagrelor
Groups:
- Ticagrelor 180mg; Ticagrelor 90mg: A total of 60 subjects will be included in this study and will be randomized in a prospective, double-blind fashion in two treatment groups: 1) 90 mg dose of ticagrelor (active comparator, standard dose); 2) 180 mg of ticagrelor (experimatal arm, loading dose).
  Ticagrelor re-load: A total of 60 subjects will be included in this study and will be randomized in a prospective, double-blind fashion in two treatment groups: 1) 90 mg dose of ticagrelor (active comparator, standard dose); 2) 180 mg of ticagrelor (experimatal arm, loading dose).
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Index (PRI) by Vasodilator-stimulated Phosphoprotein (VASP)
Description: The primary end-point of the study is the comparison in the platelet reactivity index (PRI%) determined by vasodilator-stimulated phosphoprotein (VASP) between baseline and 4-hour after dosing in each arm of treatment
Time Frame: 4 hours
Measure: Least Squares Mean (Standard Error); unit: PRI%
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Number analyzed (Participants) | 30 | 30
PRI% | 17.87 (2.1) | 23.4 (2.1)

2. Secondary Outcome: P2Y12 Reaction Units (PRU) Determined by VerifyNow P2Y12
Description: Secondary analysis included the differences of platelet reactivity expressed as P2Y12 reaction units (PRU) in each group using the VerifyNow P2Y12 system.
Time Frame: 4 hours
Measure: Least Squares Mean (Standard Error); unit: PRU
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Number analyzed (Participants) | 30 | 30
PRU | 16.8 (3.01) | 31.4 (5.2)

ADVERSE EVENTS:
Time Frame: Adverse events, including bleeding, bradyarrhythmias, and dyspnea, were recorded up to 24 hours after study completition
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes